CLINICAL TRIAL: NCT05001763
Title: A Randomized Controlled Clinical Trial of Prucaloprude Succinate in Promoting the Recovery of Intestinal Function After Robot-assisted Laparoscopic Radical Cystectomy and Urinary Diversion
Brief Title: Prucalopride for Postoperative Ileus in Patients Undergoing Robot-assisted Laparoscopic Radical Cystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUNU-UC-101
Record Dates: First submitted 2021-07-25; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Ileus; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Glucose, 2mg, tablet.
  Interventions: Drug: Placebo
- Prucalopride (Experimental): Prucalopride, 2mg, tablet. First given 2 days before surgery beginning on POD 1, until defecation or for a maximum of 7 days of postoperative treatment.
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — Prucalopride, 2mg, tablet. First given 2 days before surgery beginning on POD 1, until defecation or for a maximum of 7 days of postoperative treatment
  Other Names: Resolor
  Arms: Prucalopride
Drug: Placebo — Glucose, 2mg, tablet.
  Arms: Placebo

SUMMARY:
The first purpose is to determine whether prucalopride can promote the recovery of intestinal function after robot-assisted laparoscopic radical cystectomy and urinary diversion.

The secondary objectives is to speed up postoperative ventilation, defecation, reduce the time of first solid food tolerance, reduce postoperative hospital stay, reduce the incidence of readmission due to intestinal obstruction and the incidence of complications within 180 days.

DETAILED DESCRIPTION:
The incidence of bladder cancer is getting higher and higher. 30% of them are myometrial invasive bladder cancer, which requires radical cystectomy. This operation is more traumatic, because it involves many physiological structures, and there will be many postoperative complications, of which intestinal complications are the most common. The main manifestation is postoperative ileus (POI).

At present, one is chewing gum after surgery, and the other is the Avimopan, which is recognized as the method to promote intestinal recovery after operation. Avimopan is a peripheral μ-opioid receptor antagonist, which can improve intestinal dysfunction. Because Avimopan has not been widely used in China, its clinical application is limited. It is reported that prucalopride may be one of the methods to promote the recovery of intestinal motility after operation. Prucalopride, an alternative to benzamide, has selective 5-HT4 agonist activity and has previously been shown to significantly improve intestinal motility and transport. The drug was well tolerated and there was no obvious adverse reaction. In addition, prucalopride has been approved in Europe and America for symptomatic treatment of chronic constipation in women whose laxatives do not provide adequate relief. However, its perioperative use in radical cystectomy has not been tested. This study will test the ability and safety of prucalopride to promote the recovery of postoperative intestinal function 2 days before radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are prepared to undergo robot-assisted laparoscopic radical cystectomy + urinary diversion due to bladder tumor;
2. urinary diversion: ileal cystectomy or orthotopic neobladder;
3. age ≥ 18 years old and ≤ 80 years old;
4. ECOG score ≤ 1;
5. important laboratory indicators meet:

   1. Blood routine test: neutrophil count ≥ 1.5 × 109 g / L, leukocyte count ≥ 4.0 × 109 × 10 ~ 9/L, platelet count ≥ 100 × 109 / L, hemoglobin ≥ 9 g /dl
   2. Electrolytes: 135mmol/L ≤ serum sodium ≤ 145mmol/L , 2.25mmol/L ≤ serum calcium ≤ 2.75mmol/l, 3.5mmolexL ≤ serum potassium ≤ 5.5mmo/L; Liver function index: glutamic pyruvic transaminase (ALT) and aspartate oxaloacetic transaminase (AST) ≤ 2.5 times the upper limit of normal value (ULN), total bilirubin TBIL ≤ 1.5 × ULN;

   d. Renal function: serum creatinine ≤ 21. 5 × ULN, eGFR ≥ 30 mL / min; e. Coagulation function: international standardized ratio (INR) < 1.5. f. The left ventricular ejection fraction ((LVEF)) was 50%;
6. The drugs that affected the observation of this experiment were not used one week before the selection. Atropine drugs; P-glycoprotein inhibitors: ketoconazole, verapamil, cyclosporine A, quinidine; erythromycin;
7. Have good defecation habits, which is defecating more than 3 times a week;
8. Have no previous intestinal surgery and no history of other tumors.
9. The subjects voluntarily participated, and the subjects themselves must sign an informed consent form (ICF), to show that they understand the purpose and procedures of this study, and are willing to participate in the study. Subjects must be willing and comply with the prohibitions and restrictions set out in the study program.

Exclusion Criteria:

1. Patients who cannot tolerate radical cystectomy,
2. patients with myometrial invasive urothelial carcinoma with distant metastasis (abdominal CT scan + enhancement, chest CT scan, ECT- bone scan, PET-CT, MRI, etc.).
3. uncontrollable concomitant diseases, including, but not limited to, persistent infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, arrhythmia, interstitial lung disease, severe chronic gastrointestinal disease associated with diarrhoea, or mental illness / social conditions, which will limit compliance with research requirements, significantly increase the risk of AE or impair the patient's ability to write informed consent.
4. Patients with the allergy or hypersensitivity of prucalopride;
5. Patients with active or symptomatic viral hepatitis or other chronic liver diseases, known to be infected with human immunodeficiency virus (HIV);
6. Active pulmonary tuberculosis;
7. Patients with severe heart, liver and kidney diseases;
8. Patients with a history of constipation, which is defined as defecation less than 3 times a week, and strenuous defecation.
9. Patients with inflammatory bowel disease (ulcerative colitis or Crohn's disease);
10. Patients with rare genetic diseases such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption shall not take prucalopride.
11. Previous operations involving intestinal, history of other tumors, history of intestinal obstruction;
12. Lack of legal capacity or limitation of legal capacity;
13. Other situations in which researchers considered it inappropriate to participate in this study.

Elimination standard

1. Those who were treated with other local or systemic that interfere this study at the same time;
2. Using other foods and drugs that interfere the tolerance judgment at the same time;
3. Violating the requirements of the study scheme, not according to the dose and course of treatment specified in the study plan;
4. Poor quality, incomplete and inaccurate of data recording;
5. Poor compliance;
6. Loss of follow-up.

Termination criteria

1. Subjects require discontinuation of research treatment;
2. Deterioration of disease;
3. Any clinical AE, laboratory examination abnormalities or concomitant diseases, according to the judgment of the researchers, continuing to participate in the study is not the greatest benefit to the subjects;
4. Serious adverse events.
5. The informed consent form can no longer be signed freely because of imprisonment or forced detention for the treatment of mental illness or somatic disease (such as infectious diseases);
6. Postoperative imagings indicate ileus;
7. At the end of treatment, the function of intestines still do not recover.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to defaecation, measured in hours, from the time the surgery ends till the first observed | up to 30 days after surgery

SECONDARY OUTCOMES:
Postoperative first passing flatus reported by the patients | up to 30 days after surgery
First solid food tolerance time | up to 30 days after surgery
Postoperative C-reactive protein(CRP) | postoperative day 1 and 3
Length of postoperative hospital stay (LOS)(days) | 30 days or until hospital discharge whichever occurs first
Incidence of readmission within 180 days | up to 180 days after surgery
Incidence of complications defined according to the Clavien-Dindo Classification within 180 days | up to 180 days after surgery
Incidence of adverse events related to drug usage | up to 7 days after drug usage
  include Diarrhoea, Flatulence, Nausea, Abdominal pain, Headaches, Menstrual disorder, Dizziness, Skeletal pain, ECG nodal arrhythmia

IPD SHARING:
Plan to Share IPD: Undecided